CLINICAL TRIAL: NCT00669539
Title: An Observational Study of Optical Correction for Strabismic Amblyopia in Children 3 to <7 Years Old
Brief Title: Observational Study of Optical Correction for Strabismic Amblyopia in Children 3 to <7 Years Old
Acronym: ATS13
Status: Completed | Type: Observational
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Other Study IDs: NEI-139; 2U10EY011751 (NIH)
Record Dates: First submitted 2008-04-28; First posted 2008-04-30 (Estimated); Results first posted 2012-05-21 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Amblyopia
Keywords: Amblyopia associated with strabismus; Refractive error
MeSH Terms: conditions — Amblyopia; Refractive Errors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Combined-Mechanism Amblyopia
- Strabismus-Only Amblyopia

SUMMARY:
This study will evaluate the effectiveness of refractive correction alone for the treatment of previously untreated strabismic or combined-mechanism amblyopia in children 3 to <7 years old with visual acuity of 20/40 to 20/400

DETAILED DESCRIPTION:
This study will evaluate the effectiveness of refractive correction alone for the treatment of previously untreated strabismic or combined-mechanism amblyopia in children 3 to <7 years old with visual acuity of 20/40 to 20/400.

A recently completed PEDIG study (ATS5) found that in 3 to < 7-year-old children with previously untreated anisometropic amblyopia, refractive correction alone improved visual acuity by 2 or more lines in 77% of the patients and amblyopia resolved in at least one third of the patients. These results supported previous observations from retrospective and pilot studies as well as Stewart et al's prospective report on 18 children with anisometropic amblyopia whose visual acuity improved after treatment with spectacle correction only.

Improvement in amblyopic eye visual acuity from treatment with optimum refractive correction in cases of anisometropic amblyopia is plausible because the refractive correction treats the underlying amblyogenic condition (i.e., uncorrected unequal refractive error) by providing retinal images of more similar clarity, size, and contrast. Elimination of the dissimilar retinal images, which may act as barriers to normal visual input, allows the amblyopic eye to receive appropriate visual stimulation. In contrast, visual acuity improvement with refractive correction alone in cases of amblyopia associated with strabismus is not expected to occur when the refractive correction does not completely eliminate the strabismus and restore fusion. In such cases, the underlying amblyogenic factor of a manifest ocular deviation remains; consequently, active cortical inhibition is presumably still present. Nonetheless, Stewart and colleagues recently reported finding gains in amblyopic eye visual acuity of children with strabismic and combined-mechanism amblyopia after a period of treatment with refractive correction alone. The PEDIG also observed this to occur in a subgroup of children with previously untreated strabismic and combined-mechanism amblyopia in a recent study. Amblyopic eye acuity improved by >= 2 lines from spectacle-corrected baseline acuity in 9 (75%; 95% CI = 43% - 95%) of the 12 patients with strabismic amblyopia and in 9 (69%, 95% CI = 39% - 91%) of the 13 patients with combined-mechanism amblyopia. Mean change from baseline to maximum improvement was 2.2 +- 1.8 and 2.6 +- 2.0 lines, respectively. These results are similar to those of Stewart and colleagues who reported visual acuity improvement averaging 3.0 lines in 16 children with strabismic amblyopia and 1.9 lines in 31 children with combined-mechanism amblyopia.

Although our results support the suggestion of Stewart et al. that strabismic amblyopia can improve with spectacle correction alone, they are not conclusive because both studies had small numbers of patients. Also, our classification of strabismus was based on alignment without refractive correction. Thus, a larger controlled study is needed to confirm or refute these findings in patients with strabismic and combined-mechanism amblyopia.

The ideal study design to answer the question of whether spectacles alone can significantly improve amblyopic eye visual acuity in strabismic children is a randomized trial with a control group who does not receive optical correction. However, most pediatric eye care providers would be reluctant to randomize esotropic children with hyperopic refractive error to a control group of no optical correction because of the likelihood of some children having accommodative esotropia, which would necessitate that hyperopic spectacles be prescribed. The number of esotropic amblyopes without an accommodative component is sufficiently few to make a randomized trial not feasible. Therefore, we have chosen to perform an observational study with a large number of children with pure strabismic and combined-mechanism amblyopia in order to evaluate the effect of refractive correction in this population of patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 3 to <7 years old
* Able to perform visual acuity testing using the ATS single-surround HOTV protocol
* Amblyopia associated with strabismus (comitant or incomitant) with or without anisometropia

  *At least one of the following criteria must be met:
  * Heterotropia at distance and/or near fixation on examination (without spectacles)
  * History of strabismus surgery (or botulinum toxin extraocular muscle injection)
  * Documented history of strabismus that is no longer present (and which in the judgment of the investigator is the cause of amblyopia)
* Visual acuity measured in each eye according to the protocol procedures that meet the following criteria:

  * Amblyopic eye 20/40 to 20/400 inclusive
  * Sound eye >=20/40
  * Inter-eye acuity difference >= 3 logMAR lines (i.e., amblyopic eye acuity at least 3 logMAR lines worse than sound eye acuity)
* No previous spectacle correction
* Refractive error meeting at least 1 of the following criteria: >= 1.00D of astigmatism in the amblyopic eye, >= 1.00D spherical equivalent anisometropia, or >= +2.00D spherical equivalent hyperopia in either eye.
* Investigator wishes to prescribe spectacles to correct refractive error
* Nystagmus per se does not exclude the patient if the above visual acuity criteria are met
* Ocular examination within 2 months prior to enrollment
* Cycloplegic refraction within 2 months prior to enrollment
* No myopia = -0.25D spherical equivalent)
* Parent understands protocol and is willing to accept treatment
* Parent has home phone (or access to phone) and is willing to be contacted by Jaeb Center staff
* Relocation outside of area of an active ATS site within next 6 months not anticipated

Exclusion Criteria:

* Prior amblyopia treatment
* Current vision therapy or orthoptics
* Ocular cause for reduced visual acuity
* Prior intraocular or refractive surgery
* Strabismus surgery planned in the 9 weeks following the Baseline Visit

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Community Sample
Sampling Method: Non-Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2008-05; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan A. Cotter, O.D., M.S., Study Chair — Southern California College of Optometry at Marshall B. Ketchum University
Locations (1):
- Southern California College of Optometry, Fullerton, California, United States

REFERENCES:
- [Result] Writing Committee for the Pediatric Eye Disease Investigator Group; Cotter SA, Foster NC, Holmes JM, Melia BM, Wallace DK, Repka MX, Tamkins SM, Kraker RT, Beck RW, Hoover DL, Crouch ER 3rd, Miller AM, Morse CL, Suh DW. Optical treatment of strabismic and combined strabismic-anisometropic amblyopia. Ophthalmology. 2012 Jan;119(1):150-8. doi: 10.1016/j.ophtha.2011.06.043. Epub 2011 Sep 29. PMID 21959371

RESULTS

PARTICIPANT FLOW:
Groups:
- Combined-Mechanism Amblyopia: Chilren with strabismus and anisometropia who were prescribed refractive error correction with spectacles. The eye with worse visual acuity was labeled the amblyopic eye; the eye with better visual acuity was labeled the fellow eye. All analyses included only 1 observation per participant.
- Strabismus-Only Amblyopia: Chilren with pure strabismus who were prescribed refractive error correction with spectacles. The eye with worse visual acuity was labeled the amblyopic eye; the eye with better visual acuity was labeled the fellow eye. All analyses included only 1 observation per participant.
Period: Overall Study
Arm/Group | Combined-Mechanism Amblyopia | Strabismus-Only Amblyopia
Started | 94 | 52
Completed | 86 (Completed defined as completing 18 week primary outcome exam) | 43 (Completed defined as completing 18 week primary outcome exam)
Not Completed | 8 | 9

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Combined-Mechanism Amblyopia | Strabismus-Only Amblyopia | Total
Number analyzed (Participants) | 94 | 52 | 146
Age, Continuous [Mean (Standard Deviation); unit: years] — Age at enrollment in years
  years | 5.1 (1.1) | 4.7 (1.0) | 4.9 (1.1)
Age, Customized [Number; unit: participants] — Age at enrollment in years
  participants
    3 to <4 years | 14 | 16 | 30
    4 to <5 years | 35 | 16 | 51
    5 to <6 years | 19 | 15 | 34
    6 to <7 years | 26 | 5 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 23 | 69
  Male | 48 | 29 | 77
Race/Ethnicity, Customized [Number; unit: participants]
  Asian | 3 | 0 | 3
  Black/Aftican American | 4 | 7 | 11
  Hispanic | 4 | 7 | 11
  White | 82 | 37 | 119
  More than one race | 0 | 1 | 1
  Unknown/not reported | 1 | 0 | 1
Distance Visual Acuity Amblyopic Eye [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured in the amblyopic eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 (best) to 20/800 (worst). Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  logMAR | 0.64 (0.24) | 0.65 (0.26) | 0.64 (0.24)
Distance Visual Acuity in Fellow Eye [Mean (Standard Deviation); unit: logMAR] — Visual acuity was measured in the fellow eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol resulting in a Snellen acuity score that can range from 20/16 (best) to 20/800 (worst). Scores were converted to log of minimum angle of resolution (logMAR) equivalents for analyses (lower logMAR value is better than higher logMAR).
  logMAR | 0.09 (0.12) | 0.16 (0.11) | 0.12 (0.12)
Interocular Difference in Distance Visual Acuity [Mean (Standard Deviation); unit: logMAR lines] — The difference between eyes in logMAR visual acuity was calculated. Larger positive values of the difference indicate better visual acuity in the fellow eye, larger negative values indicate better visual acuity in the amblyopic eye, and small values indicate similar visual acuities between the eyes.
  logMAR lines | 5.4 (2.4) | 4.9 (2.2) | 5.2 (2.3)
Spherical Equivalent Refractive Error in Amblyopic Eye [Number; unit: participants] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value in the amblyopic eye. Larger values indicate more refractive error; larger spherical equivalent values are worse than smaller values.
  participants
    0 to <+1.00 diopters (better) | 1 | 1 | 2
    +1.00 to <+2.00 diopters | 8 | 3 | 11
    +2.00 to <+3.00 diopters | 5 | 17 | 22
    +3.00 to <+4.00 diopters | 17 | 10 | 27
    >=+4.00 diopters (worse) | 63 | 21 | 84
Spherical Equivalent Refractive Error in Amblyopic Eye [Mean (Standard Deviation); unit: diopters] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value in the amblyoic eye. Larger values indicate more refractive error; larger spherical equivalent values are worse than smaller values.
  diopters | 4.65 (1.79) | 3.69 (1.74) | 4.31 (1.83)
Spherical Equivalent Refractive Error in Fellow Eye [Number; unit: participants] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value in the fellow eye. Larger values indicate more refractive error; larger spherical equivalent values are worse than smaller values.
  participants
    0 to <+1.00 diopters (better) | 11 | 1 | 12
    +1.00 to <+2.00 diopters | 24 | 5 | 29
    +2.00 to <+3.00 diopters | 32 | 17 | 49
    +3.00 to <+4.00 diopters | 9 | 12 | 21
    >=+4.00 diopters (worse) | 18 | 17 | 35
Spherical Equivalent Refractive Error in Fellow Eye [Mean (Standard Deviation); unit: diopters] — Spherical equivalent in diopters defined from cycloplegic refraction as sphere plus half the cylinder value in the fellow eye. Larger values indicate more refractive error; larger spherical equivalent values are worse than smaller values.
  diopters | 2.61 (1.60) | 3.44 (1.62) | 2.90 (1.65)
Ocular Alignment [Number; unit: participants] — Minimum ocular alignment in prism diopters at distance or near defined from the simultaneous prism and cover test. Lower values of ocular alignment are better than higher values.
  participants
    0 prism diopters (better) | 23 | 14 | 37
    1-8 prism diopters | 48 | 15 | 63
    >8 prism diopters (worse) | 23 | 23 | 46
Ocular Alignment [Mean (Standard Deviation); unit: prism diopters] — Minimum ocular alignment in prism diopters at distance or near defined from the simultaneous prism and cover test. Lower values of ocular alignment are better than higher values.
  prism diopters | 5.7 (7.0) | 11.1 (14.5) | 7.6 (10.6)

OUTCOME MEASURES:

1. Primary Outcome: Mean Amblyopic Eye Visual Acuity Improvement With Spectacles
Description: Acuity is measured in each eye using the Amblyopia Treatment Study (ATS) visual acuity testing protocol at baseline and at 18wks resulting in a Snellen acuity score that can range from 20/16 to 20/800. The score is converted to logMAR (log of min angle of resolution) for statistical analysis, and a difference between the scores is calculated. A positive difference indicates acuity was better at 18wks than at baseline; a negative difference indicates acuity was worse at 18wks than at baseline.
Time Frame: Enrollment to 18 Weeks
Population: Primary analysis includes only patients who completed the 18 week exam. No imputation was done if missed exam; analysis followed the intent to treat principle.
Measure: Mean (Standard Deviation); unit: logMAR units
Arm/Group | Combined-Mechanism Amblyopia | Strabismus-Only Amblyopia
Number analyzed (Participants) | 86 | 43
logMAR units | 2.3 (1.8) | 3.2 (1.9)

ADVERSE EVENTS:
Arm/Group | Combined-Mechanism Amblyopia | Strabismus-Only Amblyopia
Serious Adverse Events (participants affected / at risk) | 0/94 | 0/52
Other Adverse Events (participants affected / at risk) | 0/94 | 0/52

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No